CLINICAL TRIAL: NCT06010758
Title: A Randomized Clinical Trial to Investigate Two-Week Clinical Safety, Changes in Salivary Flow and pH Following Use of an Anticavity Low pH Mouthwash
Brief Title: A Two-Week Study of an Anticavity Low pH Mouthwash
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCSORC005342; CCSORC005342 (Other: Johnson & Johnson Consumer Inc.)
Record Dates: First submitted 2023-07-18; First posted 2023-08-25 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Mouth wash; Mouth rinse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Brush / Listerine Experimental Mouthwash (Experimental): After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Experimental Mouthwash twice a day.
  Interventions: Drug: Listerine Experimental Mouthwash; Drug: Colgate Cavity Protection Toothpaste
- Arm 2: Brush / Listerine Cool Mint Zero (Experimental): After brushing for 1 timed minute, participants will rinse full strength for 30 seconds with experimental mouthwash twice a day.
  Interventions: Drug: Colgate Cavity Protection Toothpaste; Other: Listerine Cool Mint Zero
- Arm 3: Brush / Listerine Total Care Zero (Experimental): After brushing for 1 timed minute, participants will rinse full strength for 1 minute with experimental mouthwash twice a day.
  Interventions: Drug: Colgate Cavity Protection Toothpaste; Drug: Listerine Total Care Zero
- Arm 4: Brush only (Other): Participants will brush their teeth using a soft bristled toothbrush and Colgate Cavity Protection Toothpaste twice daily for 1 timed minute and then rinse with water for 1 minute.
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Listerine Experimental Mouthwash — After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Experimental Mouthwash twice a day, morning and night.
  Arms: Arm 1: Brush / Listerine Experimental Mouthwash
Drug: Colgate Cavity Protection Toothpaste — Participants will brush twice daily for 1 timed minute with Colgate Cavity Protection toothpaste.
Drug: Listerine Total Care Zero — After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Total Care Zero mouthwash twice a day, morning and night.
  Arms: Arm 3: Brush / Listerine Total Care Zero
Other: Listerine Cool Mint Zero — After brushing for 1 timed minute, participants will rinse full strength for 30 seconds with Listerine Cool Mint Zero mouthwash twice a day, morning and night.
  Arms: Arm 2: Brush / Listerine Cool Mint Zero

SUMMARY:
The purpose of this clinical trial is to evaluate the oral tolerance of a new, experimental mouthwash compared to two mouth rinse formulations, which are already marketed, as well as compared to a tooth brushing only control group.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the clinical trial (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical trial) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the participant (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Able to read and understand the local language (participant is capable of reading the documents)
* Adequate oral hygiene (that is, brush teeth daily and exhibit no signs of oral neglect)
* Adults, 18 years of age and older, in good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of being fully vaccinated for Coronavirus Disease 2019 (COVID-19) (adults 60 years and older)
* Negative pregnancy urine tests (females of child-bearing potential only)
* Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the clinical trial
* Resting baseline unstimulated salivary sample must be equal to or greater than 0.3 milliliters per minute (mL/min) to continue in the clinical trial
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of advanced periodontitis based on a clinical examination and discretion of the dental examiner
* Absence of fixed or removable orthodontic appliance or removable partial dentures

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouthwashes, and red food dye
* Dental prophylaxis within four weeks prior to Baseline visit
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures; Use of antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, cyclosporin A, immunostimulants/ immunomodulators during the clinical trial or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication (ibuprofen, Aspirin); oral steroids and calcium channel blockers are acceptable at the discretion of the investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, sodium fluoride with cetylpyridinium chloride (CPC), stannous fluoride, zinc or chlorhexidine digluconate containing mouthwashes and toothpastes within the four weeks prior to the Baseline exam
* Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products) specifically Cinnamyl Alcohol, Benzyl Alcohol, Citral, Citronellol, Linalool, and Limonene
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of clinical trial results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping, and e-cigarette usage
* Males with a pregnant partner or a partner who is currently trying to become pregnant
* Suspected alcohol or substance abuse (for example, amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant medical or oral condition which may interfere with a participant's participation in the clinical trial, including cancer, chronic kidney disease, chronic obstructive pulmonary disease (COPD), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) Sickle cell disease, Type 2 diabetes mellitus at the discretion of the Investigator
* Participation in any clinical trial within 30 days of Screening visit
* Diagnosed Temporo-mandibular joint dysfunction/disorder
* Participants who wear bruxing devices, dental aligners, retainers
* Participants who were previously screened and ineligible or were randomized to receive investigational product
* Participants who are related to those persons involved directly or indirectly with the conduct of this clinical trial (that is, principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Oral Tolerance as Assessed by Clinical Examinations of Oral Hard and Soft Tissues | Up to Day 14
  Oral tissue tolerance will include the assessment of the number of participants with treatment-emergent adverse events (TEAEs) and those experiencing investigational product-related AEs throughout the observational study period of 14 days. In particular, oral examinations will include clinical evaluation of soft and hard tissues, such as buccal and sublingual mucosa, tongue, hard and soft palate, gingiva, uvula, oropharynx, teeth, and dental restorations, with findings recorded in the electronic data capture (EDC) system.
Number of Participants with Adverse Events (AEs) | Up to Day 14
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participant's participation in the trial.

SECONDARY OUTCOMES:
Salivary Flow Rate | Taken at Baseline and immediately (0), and at 2.5, 5, 10, 15, and 30 minute timepoints
  Saliva samples will be collected by participants at specified timepoints. The final amount of saliva will be weighed and flow rate will be determined.
Saliva Potential of Hydrogen (pH) | Taken at Baseline and immediately (0), and at 2.5, 5, 10, 15, and 30 minute timepoints
  The pH value of saliva will be measured by placing the saliva sample onto the pH-sensitive electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.

REFERENCES:
- [Background] Lynch MC, Cortelli SC, McGuire JA, Zhang J, Ricci-Nittel D, Mordas CJ, Aquino DR, Cortelli JR. The effects of essential oil mouthrinses with or without alcohol on plaque and gingivitis: a randomized controlled clinical study. BMC Oral Health. 2018 Jan 10;18(1):6. doi: 10.1186/s12903-017-0454-6. PMID 29321067
- [Background] Cortelli SC, Cortelli JR, Shang H, McGuire JA, Charles CA. Long-term management of plaque and gingivitis using an alcohol-free essential oil containing mouthrinse: a 6-month randomized clinical trial. Am J Dent. 2013 Jun;26(3):149-55. PMID 23986962
- See also: A Randomized Clinical Trial to Investigate Two-Week Clinical Safety, Changes in Salivary Flow and pH Following Use of an Anticavity Low pH Mouthwash — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC005342&attachmentIdentifier=80eba283-d59d-4938-8fa3-a07b8aff4340&fileName=CCSORC005342_CSR_Synopsis.pdf&versionIdentifier=